CLINICAL TRIAL: NCT01238172
Title: The Men's Eating and Living (MEAL) Study: A Randomized Trial of Diet to Alter Disease Progression in Prostate Cancer Patients on Active Surveillance
Brief Title: Diet in Altering Disease Progression in Patients With Prostate Cancer on Active Surveillance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-70807; CALGB-70807; CDR0000687958 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Results first posted 2019-03-12 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Nutrition Assessment; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A - MEAL Program Intervention (Experimental): Patients will receive dietary education and telephone counseling sessions over 24 months.
  Interventions: Other: dietary education and counseling
- Arm B - Prostate Cancer Foundation Booklet (Experimental): Patients receive information about diet, nutrition, exercise and cancer. Patients also receive regularly scheduled newsletters.
  Interventions: Other: prostate cancer foundation booklet

INTERVENTIONS:
Other: dietary education and counseling
  Arms: Arm A - MEAL Program Intervention
Other: prostate cancer foundation booklet
  Arms: Arm B - Prostate Cancer Foundation Booklet

SUMMARY:
RATIONALE: Eating a diet high in vegetables may slow down disease progression in patients with prostate cancer.

PURPOSE: This randomized clinical trial is studying how well diet works in altering disease progression in patients with prostate cancer on active surveillance.

DETAILED DESCRIPTION:
CALGB 70807 is a randomized, phase III clinical trial designed to test this practical, diet-based intervention for prostate cancer in a broader clinical setting. Patients on AS will be randomized either to an intervention of centralized, telephone-based dietary counseling and structured dietary education or to a comparison control condition in which they receive the Prostate Cancer Foundation booklet. Study endpoints will include disease progression, incidence of treatment, and health-related quality of life.

OBJECTIVES:

Primary

* To determine if a telephone-based dietary intervention compared to no intervention will decrease clinical progression in AS patients.

Secondary

* To compare the incidence of active treatment (surgery, irradiation, local ablation, or androgen deprivation) in AS patients receiving dietary intervention compared to no intervention.
* To compare prostate cancer-related anxiety in AS patients receiving dietary intervention compared to no intervention.
* To compare health-related quality of life in AS patients receiving dietary intervention compared to no intervention.

OUTLINE: This is a multicenter study. Patients are stratified according to age (≤ 70 years vs > 70 years), race (black or african american vs other), and baseline prostate biopsy (0-12 months before registration vs > 12-24 months before registration). Patients are randomized to 1 of 2 treatment arms. Please see the arms section for more information.

ELIGIBILITY:
Preregistration Eligibility:

1. Histologic Documentation:

   * The initial biopsy showing diagnosis of prostate cancer should be used for the purposes of determining eligibility.
   * However, if a subsequent biopsy performed before patient enrollment shows that the patient is ineligible, he may not be enrolled to the study.
   * Eligible patients must meet all of the following criteria:

     * Biopsy-proven (consisting of ≥ 10 tissue cores) adenocarcinoma of the prostate diagnosed within 24 months prior to pre-registration
     * < 25% of biopsy tissue cores positive for cancer
     * ≤ 50% of any one biopsy tissue core positive for cancer
     * Clinical stage ≤ T2a
     * Patients who have prostate cancer with distant metastases are not eligible
   * NOTE: If a patient undergoes a transurethral resection of the prostate (TURP) for benign prostatic hyperplasia (BPH), and prostate cancer is diagnosed incidentally from the TURP specimen, eligibility for CALGB 70807 cannot be determined from the TURP specimen. However, if the patient subsequently undergoes a minimum 10-core prostate biopsy within 2 years of prostate cancer diagnosis from the TURP, and prostate cancer is detected in the biopsy specimen and meets the requirements above, the patient is eligible for this study. If prostate cancer is not detected in the biopsy specimen, the patient is not eligible.
2. Prior Treatment: Patients who have had prior treatment for prostate cancer by surgery, irradiation, local ablative (i.e. cryosurgery or high-intensity focused ultrasound) or androgen deprivation therapy are not eligible.
3. Patients who have had a history of non-cutaneous malignancy (other than nonmelanoma skin cancer) in the previous 5 years are not eligible.
4. Language: Patients must be able to read and comprehend English language text and be able to understand spoken English over the phone.
5. Life expectancy of at least 3 years
6. Patients who are currently taking vitamin supplements including lycopene and beta-carotene are eligible.
7. Patients receiving treatment with 5-alpha reductase inhibitors (e.g., finasteride, dutasteride) within 90 days prior to preregistration are not eligible. Treatment with these agents during the protocol intervention is not permitted.
8. Patients who are currently taking coumadin are not eligible.
9. Participants will be men aged 50 to 80 years.
10. For men ≤ 70 years, biopsy Gleason score ≤ 6; for men > 70 years, biopsy Gleason score ≤ (3 + 4) = 7.
11. Required Initial Laboratory Values:

    * Serum PSA < 10 ng/mL
    * NOTE: Baseline PSA for determination of eligibility must be measured after discontinuation of any 5-alpha reductase inhibitors.

Registration Eligibility:

1. Successful completion of three 24-hour dietary recalls during the run-in period.
2. Patients consuming ≥ 6 servings per day of fruits and vegetables (not including juices), as determined by the run-in dietary recalls are not eligible.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2017-11-18 (Actual); Study Completion 2019-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Kellogg Parsons, MD, MHS, Study Chair — University of California, San Diego
Locations (180):
- United States (180):
  - Fairbanks Cancer Treatment Center at Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Kaiser Permanente Medical Center - Bellflower, Bellflower, California
  - California Cancer Care, Incorporated - Greenbrae, Greenbrae, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente Medical Center - Kaiser Foundation Hospital - San Diego, San Diego, California
  - Naval Medical Center - San Diego, San Diego, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Middlesex Hospital Cancer Center, Middletown, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Cleveland Clinic Florida - Weston, Weston, Florida
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Kauai Medical Clinic, Lihue, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Oncare Hawaii, Incorporated - Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - St. Joseph Regional Medical Center, Lewiston, Idaho
  - Idaho Urologic Institute, PA, Meridian, Idaho
  - Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Bloomington Hospital Regional Cancer Institute, Bloomington, Indiana
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Wendt Regional Cancer Center at Finley Hospital, Dubuque, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - St. Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - Hays Medical Center, Hays, Kansas
  - Hutchinson Hospital Corporation, Hutchinson, Kansas
  - Kansas City Cancer Centers - West, Kansas City, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Kansas City Cancer Centers - Southwest, Overland Park, Kansas
  - Mount Carmel Regional Cancer Center, Pittsburg, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Kansas City Cancer Center - Shawnee Mission, Shawnee Mission, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - Maine Medical Center - Bramhall Campus, Portland, Maine
  - Maine Center for Cancer Medicine and Blood Disorders - Scarborough, Scarborough, Maine
  - York Hospital's Oncology Treatment Center, York Village, Maine
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - Adult and Pediatric Urology, PLLP, Sartell, Minnesota
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - Kansas City Cancer Centers - South, Kansas City, Missouri
  - Kansas City Cancer Centers - North, Kansas City, Missouri
  - Kansas City Cancer Centers - East, Lee's Summit, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Elliot Regional Cancer Center at Elliot Hospital, Manchester, New Hampshire
  - Foundation Medical Partners, Nashua, New Hampshire
  - Saint Clare's Hospital, Denville, New Jersey
  - Dizzy Gillespie Cancer Institute at Englewood Hospital and Medical Center, Englewood, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Mount Kisco Medical Group, PC, Mount Kisco, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Bay Area Hospital, Coos Bay, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Cancer Center at Phoenixville Hospital, Phoenixville, Pennsylvania
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - University Hospital - San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Auburn Regional Center for Cancer Care, Auburn, Washington
  - Overlake Cancer Center at Overlake Hospital Medical Center, Bellevue, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Cascade Cancer Center at Evergreen Hospital Medical Center, Kirkland, Washington
  - Seattle Cancer Care Alliance at EvergreenHealth, Kirkland, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Pacific Medical Center, Seattle, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - D.N. Greenwald Center, Mukwonago, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Derived] Parsons JK, Zahrieh D, Mohler JL, Paskett E, Hansel DE, Kibel AS, Liu H, Seisler DK, Natarajan L, White M, Hahn O, Taylor J, Hartman SJ, Stroup SP, Van Veldhuizen P, Hall L, Small EJ, Morris MJ, Pierce JP, Marshall J. Effect of a Behavioral Intervention to Increase Vegetable Consumption on Cancer Progression Among Men With Early-Stage Prostate Cancer: The MEAL Randomized Clinical Trial. JAMA. 2020 Jan 14;323(2):140-148. doi: 10.1001/jama.2019.20207. PMID 31935026
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 602 total patients were pre-registered, only 478 patients were deemed eligible and randomized.
Groups:
- Arm B - Prostate Cancer Foundation Booklet: Patients receive education material about diet, nutrition, exercise and cancer.
Period: Overall Study
Arm/Group | Arm A - MEAL Program Intervention | Arm B - Prostate Cancer Foundation Booklet
Started (Intention-to-treat (ITT) Cohort) | 237 | 241
Completed (modified intention-to-treat (m-ITT) Cohort) | 226 | 217
Not Completed | 11 | 24
Not completed — Ineligible: based on Eligibility Review | 2 | 5
Not completed — Ineligible: based on Central Path Review | 9 | 19

BASELINE CHARACTERISTICS:
Population: The m-ITT population included all randomized patients; however, patients who later became ineligible by eligibility review or centralized pathology review of their baseline tissue specimens were excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - MEAL Program Intervention | Arm B - Prostate Cancer Foundation Booklet | Total
Number analyzed (Participants) | 226 | 217 | 443
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (6.5) | 63.5 (6.6) | 63.6 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 226 | 217 | 443
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 9 | 15
  Black or African American | 24 | 26 | 50
  Hispanic or Latino | 9 | 7 | 16
  More than one race | 0 | 2 | 2
  Native Hawaiian or Pacific Islander | 0 | 1 | 1
  White | 186 | 171 | 357
  Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 226 | 217 | 443
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 28.7 (5.9) | 28.3 (3.7) | 28.5 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: Time to progression (TTP) was defined as the length of time from the date of random assignment to progression; patients who died from any cause without experiencing disease progression were censored at the time of death. Disease progression is defined by (a) PSA doubling time (PSADT) less than 3 years, (b) PSA above 10 at any time, or (c) Gleason score on repeat biopsy ≥ 7 for men 70 years or younger and ≥ 4+3 = 7 for men older than 70 years. For the primary analysis, TTP was analyzed using the Kaplan-Meier method; the log-rank test was used to determine superiority of the intervention arm (Arm A: MEAL Program Intervention) compared with the control arm (Arm B: Prostate Cancer Foundation Booklet).
Time Frame: Up to 2 years
Population: The primary analysis was based on the modified intention-to-treat (m-ITT) analysis population. The m-ITT population included all randomized patients; however, patients who later became ineligible by eligibility review or centralized pathology review of their baseline tissue specimens were excluded.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm A - MEAL Program Intervention | Arm B - Prostate Cancer Foundation Booklet
Number analyzed (Participants) | 226 | 217
days | 683.0 [471.0 to 733.0] | 549.0 [418.0 to 728.0]
Statistical Analysis 1: Comparison: Arm A - MEAL Program Intervention vs Arm B - Prostate Cancer Foundation Booklet; Test type: Superiority; p = 0.76, Log Rank; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.75 to 1.24]

2. Secondary Outcome: Time to Treatment: Censoring Death, Progression or Last Follow-up as Measured by Number of Events Observed
Description: Time to treatment was analyzed by the Kaplan-Meier method. For this analysis, patients who did not withdrawal from the study to pursue treatment were censored at the time of clinical progression, death, or their last follow-up visit, whichever occurred first. The number of patients who observed an event (treatment) are summarized below.
Time Frame: Up to 2 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - MEAL Program Intervention | Arm B - Prostate Cancer Foundation Booklet
Number analyzed (Participants) | 226 | 217
Participants | 3 | 2
Statistical Analysis 1: Comparison: Arm A - MEAL Program Intervention vs Arm B - Prostate Cancer Foundation Booklet; Test type: Superiority; p = 0.71, Log Rank; Hazard Ratio (HR) = 1.41, 95% CI 2-sided [0.23 to 8.41]

3. Secondary Outcome: Quality of Life (QOL) Was Measured Using Change From Baseline in Total Summary Score of Memorial Anxiety Scale for Prostate Cancer (MAX-PC) at Month 24
Description: Quality of Life (QOL) was measured using Observed Total Summary Score of Memorial Anxiety Scale for Prostate Cancer [MAX-PC] at Month 24 on a 0-108 scale, with lower scores corresponding to worse overall QOL and higher scores corresponding to better overall QOL. MAX-PC is a prostate cancer-specific measure to assess patient anxiety due to prostate cancer, PSA tests and fears of recurrence. Change from baseline to month-24 was calculated by subtracting the baseline scores from the scores at month-24. Higher scores on MAX-PC indicate better QOL
Time Frame: Up to 2 years
Population: modified ITT population: Only participants with available data on the individual study measure at baseline and 24 months were included in the analysis.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Arm A - MEAL Program Intervention | Arm B - Prostate Cancer Foundation Booklet
Number analyzed (Participants) | 150 | 140
score on a scale | 2.0 [-39.5 to 41.9] | 2.8 [-42.3 to 34.3]
Statistical Analysis 1: Comparison: Arm A - MEAL Program Intervention vs Arm B - Prostate Cancer Foundation Booklet; Test type: Superiority; p = 0.995, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Total Vegetables (Servings Per Day) Evaluated at Baseline and Month 24 Based on Dietary Recall
Description: At baseline and 24 months, participant diet including total vegetables (servings/day) was measured with a series of three separate interviews at each time point, on three-randomly selected days in a single week, using the Nutrition Data Systems for Research (NDS-R, current version 2010, University of Minnesota Nutrition Coordinating Center, University of Minnesota, Minneapolis, MN) software and nutrient database. Total vegetables were measured as the number of servings per day (range: ≥ 0), where higher values correspond to more servings per day. The within-participant change from baseline at 24 months was calculated by subtracting the baseline number of servings per day from the number of servings per day at month 24; positive values correspond to increased consumption of total vegetables.
Time Frame: Up to 2 years
Population: Participants with available data on the individual study measure at baseline and 24 months were included in the analysis
Measure: Mean (95% Confidence Interval); unit: servings per day
Arm/Group | Arm A - MEAL Program Intervention | Arm B - Prostate Cancer Foundation Booklet
Number analyzed (Participants) | 233 | 240
servings per day | 2.01 [1.75 to 2.28] | 0.37 [0.11 to 0.62]
Statistical Analysis 1: Comparison: Arm A - MEAL Program Intervention vs Arm B - Prostate Cancer Foundation Booklet; Test type: Superiority; p < 0.001, t-test, 2 sided; Two-sided

ADVERSE EVENTS:
Time Frame: Adverse events were not collected for this study.
Description: Adverse events were not collected for this study.
Arm/Group | Arm A - MEAL Program Intervention | Arm B - Prostate Cancer Foundation Booklet
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/72/NCT01238172/Prot_SAP_000.pdf